CLINICAL TRIAL: NCT03019419
Title: Perampanel for Sporadic Amyotrophic Lateral Sclerosis (ALS): A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 2 Trials
Brief Title: Perampanel for Sporadic Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tokyo Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A2016-J000-001
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: ALS
Keywords: sporadic ALS; perampanel
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perampanel 4mg (Experimental): Once daily 4mg of perampanel with dose-escalation tolerable from 2mg to 4mg for 48 weeks
  Interventions: Drug: Perampanel
- Perampanel 8mg (Experimental): Once daily 8mg of perampanel with dose-escalation tolerable from 2mg to 8mg for 48 weeks
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): Once daily placebo for control for 48 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Perampanel — 4mg/d or 8mg/d
  Other Names: non-competitive AMAP antagonist
  Arms: Perampanel 4mg; Perampanel 8mg
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
To investigate the safety and the efficacy of perampanel in patients with sporadic amyotrophic lateral sclerosis

DETAILED DESCRIPTION:
To evaluate the effect of peramanel for 48 weeks on progression of disease in subjects with ALS, as measured by ALS Functional Rating Scale-Revised (ALSFRS-R)

ELIGIBILITY:
[Eligibility Criteria for Interim Registration]

* Patients who are able to submit written informed consent. If patients are duly capable of study consent but are unable to sign by themselves due to aggravation of disease condition, written informed consent can be obtained from a legally authorized representative who can sign on behalf of the patients after confirming the patients' agreement to study participation.
* Patients who are male or female aged 40 years to 78 years at the time of obtaining informed consent
* Patients who have clinically definite ALS, clinically probable ALS, or clinically probable-laboratory supported ALS as specified in the revised El Escorial Airlie House diagnostic criteria.
* The sum of the 3 respiratory items of the ALSFRS-R must total 12 points or more
* Patients within 2-year elapsed time period from disease onset at the time of obtaining informed consent
* Patients who can visit study site for out-patient treatment

[Eligibility Criteria for Registration]

Subjects who meet the following criteria in addition to the inclusion criteria for the interim registration

* The progression on score of ALSFRS-R during 12 weeks of observation period must be between -2 and -5
* Patients who has not initiated newly introduced riluzole therapy after starting the observation period. Or those who has not received dose escalation or resumed administration of riluzole therapy after previous down titration or discontinuation
* Patients who has not initiated newly introduced edaravone therapy after starting the observation period
* Patients who are judged to be eligible for continuation of the study by the investigators

[Exclusion Criteria]

* Patients who underwent tracheostomy.
* Patients who experienced non-invasive positive pressure ventilation.
* Patients whose percent-predicted forced vital capacity (%FVC) is ≤80%.
* Patients with progressive bulbar palsy type.
* Patients with cognitive impairment, severe disease in the renal, cardiovascular, or hematological system.
* Patients with hepatic disease.
* Patients with malignant tumor.
* Pregnant women or women with a possibility of becoming pregnant.
* Patients who participated in another clinical study within 12 weeks before starting the observation period.
* Patients who has initiated perampanel therapy in the past or at present.
* Patients who are judged to be ineligible for study entry by the investigators.

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change in ALS Functional rating scale | 48 weeks

SECONDARY OUTCOMES:
Change in ALS Functional rating scale | 12, 24, 36, and 48 weeks
Manual Muscle Test | 12, 24, 36, and 48 weeks
Percent-predicted forced vital capacity | 12, 24, 36, and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Haga, Study Director — The University of Tokyo Hospital
Locations (12):
- Japan (12):
  - Kitasato University East Hospital, Kanagawa
  - Kumamoto Saishunso National Hospital, Kumamoto
  - Nagoya University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Shiga University of Medical Science Hospital, Shiga
  - Tokyo Medical University, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Neurological Hospital, Tokyo
  - University of Tsukuba Hospital, Tsukuba
  - Yamaguchi University Hospital, Yamaguchi

IPD SHARING:
Plan to Share IPD: No